CLINICAL TRIAL: NCT01973153
Title: The Added Value of Telephone Follow Up and Home Visits in Helping Children to Grow Up Healthy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Connecticut Children's Medical Center (Other)
Collaborators: Community Health Network (Other)
Responsible Party: Principal Investigator, Christine M Trapp, MD, Principal Investigator, Connecticut Children's Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHNCT-012
Record Dates: First submitted 2013-10-25; First posted 2013-10-31 (Estimated); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Obesity
Keywords: Obesity prevention; Weight management; Motivational Interviewing
MeSH Terms: conditions — Obesity | interventions — Bone Density; House Calls; Home Care Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Brief Motivational Counseling (BMC) (Active Comparator): 3-5 minute BMC delivered by clinicians and nurses at well, sick, and WIC visits with the goal of reducing obesogenic behaviors. During BMC, the medical team facilitates the selection of a specific goal (i.e., reduce sugar sweetened beverage consumption) that is meaningful to the mother and teaches the mother simple behavioral strategies.
  Interventions: Behavioral: Brief Motivational Counseling (BMC)
- Brief Motivational Counseling Plus Phone Calls (BMC+Phone) (Active Comparator): BMC as described above that is supplemented by monthly telephone contacts with community health workers designed to identify and overcome barriers to goal progress.
  Interventions: Behavioral: Brief Motivational Counseling (BMC); Behavioral: Brief Motivational Counseling Plus Phone Calls (BMC + Phone)
- Brief Motivational Counseling Plus Home Visits (BMC+Home) (Active Comparator): BMC as described above that is supplemented by monthly home visits with community health workers designed to identify and overcome barriers to goal progress.
  Interventions: Behavioral: Brief Motivational Counseling (BMC); Behavioral: Brief Motivational Counseling Plus Home Visits (BMC + Home)

INTERVENTIONS:
Behavioral: Brief Motivational Counseling (BMC) — 3-5 minute BMC delivered by clinicians and nurses at well, sick, and WIC visits with the goal of reducing obesogenic behaviors. During BMC, the medical team facilitates the selection of a specific goal (i.e., reduce sugar sweetened beverage consumption) that is meaningful to the mother and teaches the mother simple behavioral strategies.
Behavioral: Brief Motivational Counseling Plus Phone Calls (BMC + Phone) — BMC as described above that is supplemented by monthly telephone contacts with community health workers designed to identify and overcome barriers to goal progress.
  Arms: Brief Motivational Counseling Plus Phone Calls (BMC+Phone)
Behavioral: Brief Motivational Counseling Plus Home Visits (BMC + Home) — BMC as described above that is supplemented by monthly home visits with community health workers designed to identify and overcome barriers to goal progress.
  Arms: Brief Motivational Counseling Plus Home Visits (BMC+Home)

SUMMARY:
Leading medical organizations have called on primary care pediatricians to take a central role in the prevention of childhood obesity. Weight counseling typically has not been incorporated into routine pediatric practice due to time and training constraints. Brief interventions with simple behavior change messages are needed to reach high-risk children, particularly Latino and Black children who are disproportionately affected by obesity and related comorbidities. Steps to Growing Up Healthy (Added Value) is a randomized controlled trial testing the efficacy of brief motivational counseling (BMC) delivered by primary care clinicians and the added value of supplementing BMC with monthly contact by community health workers (CHW) in the prevention/reversal of obesity in Latino and Black children ages 2-4 years old. Mother-child dyads (targeted n=150) are recruited for this 12-month randomized trial at an inner-city pediatric primary care clinic and randomized to: 1) BMC delivered by clinicians and nurses at well, sick, and WIC visits with the goal of reducing obesogenic behaviors (BMC); 2) BMC plus monthly phone calls by a CHW (BMC+Phone); or 3) BMC plus monthly home visits by a CHW (BMC+Home). During BMC, the medical team facilitates the selection of a specific goal (i.e., reduce sugar sweetened beverage consumption) that is meaningful to the mother and teaches the mother simple behavioral strategies. Monthly contacts with CHWs are designed to identify and overcome barriers to goal progress. Dyads are assessed at baseline and 12 months and the primary outcome is change in the child's BMI percentile. We hypothesize that BMC+Phone and BMC+Home will produce greater reductions in BMI percentiles than BMC alone and that BMC+Home will produce greater reductions in BMI percentiles than BMC+Phone.

ELIGIBILITY:
Inclusion Criteria:

* Child is 2-4 years old
* Latino or Black descent by maternal report
* Receiving services through the Special Supplemental Nutrition Program for Women, Infants, and Children (WIC)

Exclusion Criteria:

* Mother is younger than 18 years old
* Dad does not live in the Greater Hartford area or if they have plans to move out of the area in the next 12 months
* Child or mother has special needs (dietary, physical, and/or emotional) that would make the intervention inappropriate (e.g. failure to thrive, type 1 diabetes, cystic fibrosis)

Ages: 2 Years to 50 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in BMI Percentile | baseline and 12 months
  BMI Percentile calculated using the 2000 revised CDC/NCH growth charts for the United States

CONTACTS AND LOCATIONS:
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States

REFERENCES:
- [Derived] Gorin AA, Wiley J, Ohannessian CM, Hernandez D, Grant A, Cloutier MM. Steps to Growing Up Healthy: a pediatric primary care based obesity prevention program for young children. BMC Public Health. 2014 Jan 23;14:72. doi: 10.1186/1471-2458-14-72. PMID 24456698